CLINICAL TRIAL: NCT01957813
Title: Development and Evaluation of an Intervention to Increase Family Planning Use Among Female Sex Workers in Kenya
Brief Title: Evaluation of a Peer Education Program to Promote Family Planning Among Female Sex Workers in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Gold Star Kenya (GSKenya) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10285
Record Dates: First submitted 2013-09-04; First posted 2013-10-08 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: APHIA AIDS, Population and Health Integrated Assistance; DIC Drop-in center; DMPA depot medroxyprogesterone acetate; DRH Division of Reproductive Health; FAIR Family AIDS Initiative Response; FHOK Family Health Options Kenya; FP Family planning; FGD Focus group discussion; FSW Female sex worker; GSKenya Gold Star Kenya; HTC HIV testing and counseling; HIV Human Immunodeficiency Virus; KNASP Kenya National AIDS Strategic Plan; MARPS Most at-risk populations; MoPHS Ministry of Public Health and Sanitation; MMS Ministry of Medical Services; NASCOP National AIDS and STI Control Program; RH Reproductive health; SRH Sexual and reproductive health; STI Sexually transmitted infection; USAID United States Agency for International Development
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Health Services (Other): Service currently being provided to FSW in Naivasha include peer education and health services delivered through a drop-in center (DIC) staff by a counselor and a nurse. For peer education, there are six modules that the peer educators walk all peers through with sessions being held once a week.
  Interventions: Other: Standard Health Services
- LifeStyle Counseling (Experimental): A package of enhancements to the current package of services delivered to FSW will be implemented and evaluated.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Peer educators will be trained using existing materials to deliver accurate messaging on FP/dual method use, during individual encounters and in group sessions.
  Screening for unmet FP need in DICs Providing job aids to FP counselors Expanding FP methods with intra-uterine contraceptive devices (IUCD) and implants Time change in DIC hours of operation
  Arms: LifeStyle Counseling
Other: Standard Health Services — Peer education and health services
  Arms: Standard Health Services

SUMMARY:
-Purpose: To develop and evaluate an intervention designed to improve consistent contraceptive use and dual method use in particular, among female sex workers (FSWs) in Rift Valley Province in Kenya.

Design: A qualitative descriptive study will be conducted to develop the intervention. A quasi-experimental, non-randomized, two-group, pre-/post-intervention design will be used to evaluate the intervention.

Study Population: FSWs living in Naivasha, Gilgil, and Nanyuki, Rift Valley Province.

Study Duration: Phase I - 3 months Phase II - 12 months Objectives: Develop an intervention designed to increase contraceptive use among FSWs by incorporating formative data and behavioral theory and by involving the target audience and service providers in the development of the intervention.

Examine the effectiveness of the intervention at increasing non-barrier modern contraceptive use and dual method use among FSWs.

Assess the feasibility and acceptability of the intervention, on the parts of both the clients (FSW) and service providers.

Estimate the unit cost to provide these services to one client. Study Site: Rift Valley Province, Kenya

DETAILED DESCRIPTION:
The goal of this study is to develop and evaluate a theory-based intervention that could be incorporated into routine health services to improve the sexual and reproductive health of women who engage in sex work if demonstrated to be effective. To accomplish this goal, the study will be conducted in two phases. During the first phase of the study, FSWs and service providers in the study sites will assist in the design of the intervention, in an effort to increase the likelihood that it will be accepted, feasible, and effective. Brief formative research will be conducted with FSWs and service providers, followed by working group meetings with self-selected FSWs, service providers, and GSKenya representatives who will review data and work with study investigators and/or their designees to design the intervention. During the second phase of this study, the intervention will be implemented and evaluated.

The study is planned for two sites within Rift Valley Province, Kenya. The first "site" is comprised of two adjacent towns, Naivasha and Gilgil. The town of Nanyuki will serve as the second site.

Based on findings from the formative phase of this study, and on observations and feedback from providers, a package of enhancements to the current package of services delivered to FSW will be implemented and evaluated.

* Family Planning (FP) Messaging for peer educators and informational materials material - Peer educators will be trained using existing materials to deliver accurate messaging on FP/dual method use, during individual encounters and in group sessions.
* Screening for unmet FP need in drop-in centers - Integration of FP needs screening in the service delivery points will increase the number of FSW accessing FP. This will be done through sensitization of service providers and provision of a brief job aid that can be used to screening clients for unmet need, including unmet need for dual method use.
* Providers FP counseling job aid - The AIDS, Population and Health Integrated Assistance (APHIA) Plus project will adapt the existing Balanced Counseling Strategy Plus: A Toolkit for Family Planning Service Providers Working in High HIV/Sexually Transmitted Infection (STI) Prevalence Settings for providers to use within the context of the DICs and in referral sites in the catchment area.
* Commodities - increasing method mix - The methods that will be available to all women attending services at the DIC will be expanded. In addition to the current oral contraceptive pills, DMPA, male and female condoms, both the intra-uterine contraceptive devices (IUCD) and implants will be added to the mix of methods available.

Hours of DIC operation - Based on findings from the formative phase of the study, the hours of operation for DICs will be extended into the late evening hours to accommodate the schedules of FSW.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a FSW. For the purposes of this study, a FSW is defined as a woman who is sexually active and reports receiving money or goods in exchange for sex in the last 6 months as part of her source of income/livelihood.
* Is between the ages of 16 and 49 years
* Provides oral informed consent

Exclusion Criteria:

-

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 719 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
Dual Method Contraceptive Use | 6 months
  Dual method use is the use of a non-condom modern method in the past month plus reported use of a condom (male or female) at last sex with both paying and non-paying partner (if applicable).

SECONDARY OUTCOMES:
Acceptability and Feasibility among providers | 6 months
  Provider acceptability is a measure of the proportion of providers at baseline and post-intervention who are strongly in favor of providing FP services to FSWs in other DICs in Kenya and the proportion of providers who are satisfied with the training and support they received to provide FP services.
  Feasibility is a measure of the proportion of providers at baseline and post-intervention who agree or strongly agree that the FP needs of FSWs receiving services at the DIC are met. In addition, there will be a measure of the proportion of providers who report that they did not have to turn a FSW client away because they were too busy or they did not have the supplies they needed.
Acceptability and feasibility of intervention among Clients | 6 months
  Client acceptability will be measured by the proportion of clients post-intervention reporting that they are satisfied or very satisfied with the services they received at the DIC and from Peer Educators, as well as a comparison of reported service convenience and satisfaction with DIC services.
  Feasibility will be measured among clients who reported receiving FP methods or services from the DIC and we will compare reported service convenience and satisfaction with DIC services at baseline and post-intervention
Acceptability and feasibility of Intervention among Peer Educators (PE) | 6 months
  Acceptability is a measure of the the proportion of PEs who are satisfied with the training and support they received to provide FP education and counseling to FSWs in the intervention site at 6 months post-intervention and the proportion of PEs reporting satisfaction with their work and motivation to perform their responsibilities as a PE.
  Feasibility is the proportion of PEs reporting that they found their responsibilities as a PE easily manageable and would choose to be a PE again.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dulli, PhD, MHS, Principal Investigator — FHI 360
Locations (2):
- Kenya (2):
  - APHIA Plus HIV Prevention Drop-in Centers, Naivasha, Rift Valley Province
  - APHIA Plus HIV Prevention Drop-in Centers, Nanyuki, Rift Valley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dulli L, Field S, Masaba R, Ndiritu J. Addressing broader reproductive health needs of female sex workers through integrated family planning/ HIV prevention services: A non-randomized trial of a health-services intervention designed to improve uptake of family planning services in Kenya. PLoS One. 2019 Jul 24;14(7):e0219813. doi: 10.1371/journal.pone.0219813. eCollection 2019. PMID 31339919